CLINICAL TRIAL: NCT06761430
Title: A PRE-MARKET, DUBLE CENTER, INTERNATIONAL, ONE-ARM, CONTROLLED, PROSPECTIVE CLINICAL INVESTIGATION ASSESSING THE SAFETY OF A CLASS IIb MEDICAL DEVICE (CLEARPLASMA™) FOR THE TREATMENT OF PATIENTS WITH ACUTE UPPER GASTROINTESTINAL HEMORRHAGE"
Brief Title: Evaluation of ClearPlasma in Patients With Upper Gastrointestinal Bleeding.
Acronym: CLearPlasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PlasFree Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLas-Free 2019-10-30_007461; DGDMF/P/I.5.I.M.2/2019/1319 (Registry Identifier: ITALIAN MOH); MOH_2019-10-30_007461 (Registry Identifier: Israeli MOH)
Record Dates: First submitted 2024-12-11; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Upper Gastrointestinal Bleeding (UGIB)
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: To assess the safety of a one-time infusion of up to two units of PDP obtained through filtration with ClearPlasma in the reduction of re-bleeding in Patients presenting with acute upper gastrointestinal hemorrhage
Masking Description: in this study there is no Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- One-time infusion of up to two units of PDP obtained through filtration with ClearPlasma (Experimental): To assess the safety of a one-time infusion of up to two units of Plasminogen depleted Plasma (PDP) obtained through filtration with ClearPlasma in Patients with acute upper gastrointestinal bleeding.
  Interventions: Device: ClearPlasma

INTERVENTIONS:
Device: ClearPlasma — ClearPlasmais an extra-corporeal plasma filtration device, designed to specifically extract plasminogen, a protein that drives fibrinolysis, from up to 250 mL of plasma. ClearPlasmaTM is a non-pyrogenic, sterile, single-use medical device.

SUMMARY:
Upper gastrointestinal hemorrhage (UGIH) is one of the most common gastrointestinal emergencies, and is associated with significant morbidity and mortality. Plas-Free aims to evaluate ClearPlasma safety in patients with UGIH.

DETAILED DESCRIPTION:
Upper gastrointestinal hemorrhage (UGIH) is one of the most common gastrointestinal emergencies, and is associated with significant morbidity and mortality. Acute upper gastrointestinal hemorrhage (AUGIH) management guidelines call for aggressive hemodynamic resuscitation, prevention and treatment of complications and treatment of bleeding, which generally includes endoscopic intervention and transfusion of appropriate blood components. However, in many cases, spontaneous hyperfibrinolysis occurs, jeopardizing pharmacological control of AUGIH. Antifibrinolytic drugs are considered effective in counteracting hyperfibrinolysis, but are associated with various side effects, such as neurotoxicity and accelerated fibrinolysis upon prolonged use.

Fibrin clot breakdown is actively mediated by plasmin, a serine protease which cleaves fibrin. Administration of plasma depleted of plasminogen, the precursor of plasmin, may shift the balance towards coagulation.

PlasFree Ltd. has developed ClearPlasma, a single-use, extracorporeal plasma filtration device which extracts plasminogen from plasma to reduce fibrinolysis. The resulting plasminogen-depleted plasma (PDP) is expected to reduce risk of fibrinolysis and re-bleeding in Patients undergoing plasma transfusions.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged ≥ 18 and ≤ 80 years old. 2. Patients presenting with acute upper gastrointestinal hemorrhage (> 0.5 L), diagnosed by presence of blood in gastric lavage, hematemesis or melena within no longer than 24 h before enrolment.

  3. Patients presenting with acute upper gastrointestinal hemorrhage (< 24 h) for which fresh frozen plasma (FFP) has been ordered.

  4. Patients understanding the nature of the study and providing their informed consent to participation.

  5. Patients willing and able to attend the follow-up visits and procedures foreseen by the study protocol.

Exclusion Criteria:

Patients who underwent a plasma infusion in the 30 days before enrolment. 2. Patients in a life-threatening condition at the time of enrolment (i.e. heart attack).

3. Patients who are hemodynamically unstable and required pressor administration at the time of enrolment (i.e. with hypovolemic shock) 4. Patients with known renal failure (creatinine clearance < 30 mL/min) at the time of enrolment.

5. Patients suffering from Hemophilia A or B. 6. Patients suffering from venous and arterial thromboembolic events within 3 months before the enrolment.

7. Patients with increased risk of blood clotting, according to Investigator's judgement.

8. Patients with fluid accumulation in the brain at the time of enrolment. 9. Patients with retinal thrombosis at the time of enrolment. 10. Patients with measured body weight < 45 kg at the time of enrolment. 11. Patients with history of allergic reaction to plasma, polyethersyplone or polycarbonate.

12. Patients suffering from IgA deficiency at the time of enrolment. 13. Patients with history of hemorrhage while on anticoagulant treatment (warfarin, apixaban, rivaroxaban, dabigatran, low molecular weight heparin).

14. Patients identified by the Investigator to have any underlying medical Clinicalconditions that may preclude conduct of study procedure (i.e. making the administration of study treatment hazardous) or obscure the interpretation of safety objectives.

15. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.

16. Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation and for 3 months later.

17. Female Patients of childbearing age (less than 12 months after the last menstrual cycle) who do not use adequate contraception *.Methods at low risk of contraceptive failure (less than 1% per year) when used consistently, including: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intra-uterine devices.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Number of severe adverse events | 30 days
  Number of severe adverse events (SAE) and/or adverse events (AE) compared to the gold standard.

SECONDARY OUTCOMES:
Thromboembolic Events | 30 days
  Venous thromboembolism (VTE) and/ or deep vein thrombosis (DVT) and/or pulmonary embolism (PE) compared to the gold standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Area Medicina D'Urgenza e Pronto Soccorso Fondazione Policlinico Universitario A. Gemelli IRCCS Università Cattolica del Sacro Cuore Largo A. Gemelli, 800168 -, Rome, Italy

IPD SHARING:
Plan to Share IPD: No